CLINICAL TRIAL: NCT06552247
Title: Validation Study of an Artificial Algorithm for Glaucoma Detection in an African Population
Brief Title: Glaucoma Algorithm Validation Study in African Population - the MAGIC Study
Acronym: MAGIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário Lisboa Norte (Other)
Collaborators: Dr. Agarwal's Eye Hospital (Industry)
Responsible Party: Principal Investigator, Luis Abegao Pinto, Co-principal investigator, Centro Hospitalar Universitário Lisboa Norte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Collaboration Mozambique 2
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma; Diabetic Retinopathy
Keywords: Artificial Intelligence; Validation; Screening
MeSH Terms: conditions — Glaucoma; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Single arm. Consecutive patients in a general ophthalmology consultation will be offered intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-based fundus picture screening (Experimental): Volunteers will performed a full study visit as part of their regular Ophthalmology assessment. This will include a fundus picture, an Optic-disc entered OCT, a Visual Field exam and a clinical examination by a clinical expert.
  Fundus picture will be assessed by an AI algorithm (G-Risk) and labelled with referral vs non-referrable and compared with the clinical gold standard
  Interventions: Diagnostic Test: Fundus Picture AI testing

INTERVENTIONS:
Diagnostic Test: Fundus Picture AI testing — G-Risk AI algorithm will assess the optic disc centered fundus picture and determine whether or not there is a need for referrable based on a pre-determined threshold (>=0.73)

SUMMARY:
Artificial Intelligence (AI) algorithms require validation in a variety of populations to ensure widespread clinical applicability. In Ophthalmology, AI algorithms are reaching maturity in diagnosis such as diabetic retinopathy and glaucoma. Higher-at-risk subjects of African descent are nevertheless usually under-represented in training datasets and therefore unclear about representativity.

A small scale validation study in consecutive patients in a large Eyesore unit in Mozambique will be performed to determine the diagnostic ability of these AI softwares in this population

DETAILED DESCRIPTION:
Artificial Intelligence (AI) algorithm's are the next frontier in medical management, usually meant to improve diagnostic capabilities and to optimize the existing resources. They are particularly relevant in settings where there is a lack of specialised Human Resources such as physicians.

Ensuring these algorithms can be used in a wide population is therefore crucial to clinical implementation. Validation studies in specific segments of populations are needed to ensure all patients are represented and the results are therefore reliable. Higher-at-risk subjects of African descent are nevertheless usually under-represented in training datasets and therefore unclear about representativity.

A pilot study for validation of an AI algorithm for Glaucoma and Diabetic Retinopathy will be done for the MONA G-RISK® and diabetic retinopathy. Consecutive patients from a large Eye Unit in Mozambique's capital will be screened using these AI algorithms and validated using clinical standard as ground truth.

ELIGIBILITY:
Inclusion Criteria:

* subjects age above 18 years old presenting at the Eye Unit
* willingness to sign an informed consent for the screening process

Exclusion Criteria:

* none
* Poor quality in screening image will be included in the intention to treat analysis, but excluded from the diagnostic comparator outcome.
* Patients with a known glaucoma diagnosis will not be excluded from the screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-14 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic agreement between referring decision and reading center decision | Duration of the study - 3 weeks
  Level of agreement will be done between referring decision and the ground truth as assessed by the reading center (normal, glaucoma suspect; definitive glaucoma). All subjects from both centers (referred and non-referred) will be reviewed.
  For a primary outcome analysis, the middle category (glaucoma suspect) will be pooled together with the normal diagnosis

SECONDARY OUTCOMES:
Level of agreement (in %) between AI-risk score and human-based assessment of disease severity | After the study - 6 months
  Reading center risk score of disease severity (ranked from 0 to 100) will be compared to the AI-based disease score. This will be done separately in each of the 3 categories (normal; glaucoma suspect; glaucoma). Analysis of this score would help refine clinical risk (high risk vs low risk patients) of each category. Exploratory analysis will be made to determine the added value of including this risk score in refining AI-based referral

CONTACTS AND LOCATIONS:
Overall Officials: Joana Ferreira, MD, PhD, Study Director — ULS Santa Maria; Amelia Buque, MD, Study Director — Dr. Agarwal Eye Hospital

IPD SHARING:
Plan to Share IPD: No